CLINICAL TRIAL: NCT05134272
Title: Infant Modified Constraint Induced Movement Therapy Paired With Neuromuscular Electrical Stimulation: a Case Series
Status: Completed | Type: Observational
Sponsor: Kathy Grinde (Other)
Responsible Party: Sponsor-Investigator, Kathy Grinde, Physical Therapist, Rehab Clinical Specialist, Children's Hospitals and Clinics of Minnesota
Organization: Children's Hospitals and Clinics of Minnesota (Other)
Other Study IDs: infantconstraint2021
Record Dates: First submitted 2021-11-08; First posted 2021-11-24 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Hemiplegia; Cerebral Palsy; Unilateral Cerebral Palsy
Keywords: infant; constraint induced movement therapy; early intervention; cerebral palsy
MeSH Terms: conditions — Hemiplegia; Cerebral Palsy | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- mCIMT plus NMES: Phase 1: Infants will receive therapy 1 hour/day, 1 day/week for 3 weeks while wearing a sock 1 hour/day. Parents will complete home program activities 1 hour/day, 6 days/week for 3 weeks.
  Phase 2:Infants will receive therapy 2 hours/day, 3 days/week for 3 weeks while wearing a splint 24 hours/day. Parents will complete home program activities 1 hour/day, 6 days/week for 3 weeks.
  Phase 3:Infants will receive therapy 1 hour/day, 1 day/week for 3 weeks while wearing a sock 1 hour/day. Parents will complete home program activities 1 hour/day, 6 days/week for 3 weeks.
  Interventions: Device: Neuromuscular electrical stimulation; Behavioral: Modified constraint induced movement therapy; Behavioral: Standard care for infant with asymmetrical hand function

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — Neuromuscular Electrical Stimulation will be applied by the therapist to infant's finger flexors and extensor for 15 min./day, 3x/week.
  Other Names: NMES
Behavioral: Modified constraint induced movement therapy — Modified CIMT will consist of constraint 24 hours/day using a splint in addition to therapy two hours/day, 3x/week for three weeks. Parents will be trained to carry over home program activities one hour/day, 6 days/week.
  Other Names: mCIMT
Behavioral: Standard care for infant with asymmetrical hand function — Infants will receive one hour of therapy, one time/week for three weeks. Parents will be trained to carry over home program activities one hour/day, 6 days/week. In addition the infant will wear a sock on their preferred hand during the hour of therapy/home program activity.

SUMMARY:
This study will compare the motor outcomes for five infants with asymmetrical hand function (AHF) who will receive two, three week episodes of standard care separated by a three week episode of mCIMT paired with Neuromuscular Electrical Stimulation. The results of this study will inform decisions on the feasibility and efficacy of the treatment for use in a larger study for infants with AHF at risk for unilateral cerebral palsy.

DETAILED DESCRIPTION:
Infants with asymmetrical hand function will participate in three consecutive phases of treatment.

The first and third phase will consist of three weeks of standard care for children with asymmetrical hand function, 1 hour/day, 1 day/week. The therapist will provide weekly coaching with the parents so they can carry over activities at home one hour/day, six days/week during this phase. In addition, a sock or mitten will be used for short term constraint during the hour of training both in the clinic with the therapist and at home with the parent.

The second phase will consist of three weeks of modified constraint induced movement therapy, 2 hours/day, 3 days/week paired with NMES, 15 minutes/day, 3 days/week. The infants will wear a soft splint on their preferred hand and forearm 24 hours/day during this phase. Parents will be trained by the therapist to carry over activities with their child at home, 1 hour/day, 6 days/week.

The children will return at chronological age of 18 months for follow up testing.

ELIGIBILITY:
Inclusion Criteria:

1. Infant is 7-10 months of age (CCA)
2. Clinical presentation of asymmetrical hand function,
3. Grade 2/5 movement in more impaired upper extremity,
4. Demonstrate potential to participate in 6 hours of therapy/week during 3 week episode of mCIMT-NMES, as determined by principal investigator,
5. Parent/guardian willing to be partners in study and participate in follow-up assessments until child is 18 months of age

Exclusion Criteria:

1. Medical or sensory condition that prevents full therapy participation (active seizures, significant visual impairment)
2. Received Botox injection to more impaired upper extremity within last 6 months,
3. NMES contraindicated (impaired skin integrity, presence of pacemaker, clotting disorder),
4. Previous UE surgery or nerve injury (brachial plexus)

Ages: 7 Months to 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with asymmetrical hand function
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in hand use based on the Hand Assessment of Infants | Baseline, week 4, week 7, week 10
  A criterion, norm referenced assessment that evaluates and measures goal directed both hand use and possible upper limb asymmetry in infants at risk of developing cerebral palsy,aged 3-12 months.

SECONDARY OUTCOMES:
Change in motor skills based on the Peabody Developmental Motor Scales-2 | Baseline, week 4, week 7, week 10, 18 months CCA
  A criterion and norm referenced test that measures fine and gross motor skill
Assisting Hand Assessment Version 4.4 | 18 months CCA
  A criterion-referenced test that measures and describes how effectively children who have unilateral disability, aged 18 months to 12 years, use their affected hand in bimanual activity performance.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy S Grinde, PT, Principal Investigator — Children's Minnesota
Locations (1):
- Children's Minnesota, Maple Grove, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No